CLINICAL TRIAL: NCT07087665
Title: Patient Satisfaction, Quality of Vision, and Quality of Life Following Treatment With WaveLight Plus LASIK
Brief Title: Patient Reported Outcomes With WaveLight Plus LASIK
Status: Enrolling by invitation | Type: Observational
Sponsor: OVO LASIK + Lens (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: ML-25-01
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Wavelight Plus — The WaveLight EX500 laser system, in conjunction with INNOVEYES Sightmap, is indicated for use in INNOVEYES Laser Assisted In-Situ Keratomileusis ("wavelight plus"1 LASIK) treatments:
  * or the reduction or elimination of myopia or myopia with astigmatism, in eyes with spherical equivalent (SE) more than -1.00 and up to -9.00 diopters (D), with up to -8.00 D of spherical component (in minus cylinder format) and up to -3.00 D of astigmatic component at the spectacle plane, based on the INNOVEYES Sightmap Measured Refraction,
  * in patients with magnitude of the spherical equivalent (SE) difference between the Manifest Refraction (MRSE) and the Sightmap measured refraction SE being less than 0.75D,
  * in patients who are 18 years of age or older, and
  * for patients with documentation of a stable manifest refraction defined as 0.5 D preoperative spherical equivalent shift over one year prior to surgery.

SUMMARY:
This study is a single-site, single-arm, prospective, observational study of subject satisfaction, quality of vision, and quality of life after bilateral LASIK surgery. Subjects will be assessed 6 months post-operatively. Clinical evaluations will include refractive outcomes, visual acuity, and administration of the adapted PROWL, QIRC, and OSDI questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and sign an approved consent form.
* Willing and able to comply with scheduled visits and other study procedures.
* Age: 18 to 37
* Myopia with or without astigmatism and MRSE within the range indications for wavelight plus (myopia up to -8 D, astigmatism up to -3.0 D, S.E. more than -1.00 and up to -9.00D)
* Pre-surgery BCDVA of 20/20 (0.00 logMAR) or better in each eye.
* Stable refraction (within ± 0.50 D) as determined by manifest refraction spherical equivalent for a minimum of 12 months prior to surgery.
* Refractive target of bilateral emmetropia
* Mesopic pupil size ≥ 4.5mm
* Less than 0.75 D spherical equivalent difference between Sightmap measured refraction SE and the subjective manifest refraction (MRSE)

Exclusion Criteria:

* Subjects with a history of previous ocular surgery.
* Subjects with topographic evidence of keratoconus or ectasia.
* Pre-existing retinal or corneal pathology Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.
* Systemic disease likely to affect wound healing, such as diabetes and severe atopy.
* Any ocular disease (including uncontrolled dry eye) in which the investigator's opinion would affect the outcome of refractive surgery.
* Patients with a calculated residual stromal depth <250 µm would be excluded from the study.

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible participants will be 18 to 37 years of age and who are candidates for Wavelight Plus LASIK to correct myopia or myopic astigmatism.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects satisfied (Completely Satisfied or Very Satisfied) with vision after Wavelight Plus LASIK based on an adapted PROWL Questionnaire (Question #1 only). | 6 months postoperatively

SECONDARY OUTCOMES:
Remaining Vision quality and quality of life during daily tasks using the adapted PROWL | 6 months postoperatively
The percentage of eyes at each monocular visual acuity (VA) level (uncorrected 20/10, 20/12.5, 20/16, 20/20, 20/25). | 6 months postoperatively
The percentage of subjects at each binocular visual acuity (VA) level (uncorrected 20/10, 20/12.5, 20/16, 20/20, 20/25). | 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Lobanoff, MD, Principal Investigator — OVO LASIK + Lens
Locations (1):
- Ovo Lasik + Lens, Saint Louis Park, Minnesota, United States